CLINICAL TRIAL: NCT06462391
Title: Adapting and Piloting Acceptance and Commitment Therapy (ACT) for Severe Premenstrual Mood Symptoms: An Open-label Feasibility Study of ACT-PM
Brief Title: Adapting and Piloting Acceptance and Commitment Therapy (ACT) for Severe Premenstrual Mood Symptoms
Acronym: ACT-PM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Principal Investigator, Elisabeth Wright, Psychiatrist, Principal Investigator, Women's College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: WCH-24-001
Record Dates: First submitted 2024-05-16; First posted 2024-06-17 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Premenstrual Dysphoric Disorder; Premenstrual Exacerbation of Mood Disorder
MeSH Terms: conditions — Premenstrual Dysphoric Disorder | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: open label pilot feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (open label) (Other): all participants will be in pilot psychotherapy group
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT) Group

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) Group — Psychotherapy group (delivered virtually)

SUMMARY:
In the weeks prior to menstruation, many individuals experience mood and physical symptoms that negatively impact their quality of life and functioning. Approximately 5% of women and menstruating individuals have such severe symptoms that they meet criteria for Premenstrual Dysphoric Disorder (PMDD). Further, of those with underlying mood disorders (i.e., depression, bipolar disorder) about 60% have cyclical worsening of symptoms classified as premenstrual exacerbation (PME). Both PMDD and PME are associated with significant impairment, yet limited effective options exist to treat these conditions. In this project, the investigators will adapt and evaluate an Acceptance and Commitment Therapy (ACT) group for PMDD and PME, entitled ACT-Premenstrual (ACT-PM), delivered virtually to maximize accessibility. The investigators will examine whether ACT-PM is feasible to deliver and whether it is acceptable to group participants and those facilitating the group. The study will lay the groundwork for future research to determine if the group is effective. If effective, the intervention could be scaled up to improve quality of life and outcomes for individuals suffering from PMDD and PME.

ELIGIBILITY:
Inclusion Criteria:

* (1) diagnosed by the psychiatrist who conducted the initial assessment with either Premenstrual Dysphoric Disorder (PMDD), or a bipolar or depressive disorder where there is Premenstrual Exacerbation (PME), after 2-3 months of mood tracking using a validated evidenced based scale for premenstrual mood symptoms (McMaster Premenstrual And Mood Symptom Scale (MAC-PMSS) or similar;
* (2) have internet access and a video-enabled device;
* (3) residing in Ontario for the duration of the study, necessary because MDs and therapists who could deliver the intervention are all licensed provincially;
* (4) regular menstrual cycles (~21-35 days); and
* (5) have a regularly treating physician (e.g. psychiatrist or primary care provider).

Exclusion Criteria:

* (1) active alcohol or substance use disorder in the previous 12 months;
* (2) active suicidal ideation, mania, psychosis, or violence;
* (3) current pregnancy or planning a pregnancy during the duration of the study
* (4) inability to complete group and/or study measures in English, necessary as the pilot group is only available in English at this time.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment and enrollment: number of participants referred | Screening and baseline
  Tracking to see how many referrals are made to the study
Feasibility of recruitment and enrollment: number of participants eligible | Screening and baseline
  Tracking number of participants that were eligible out of the number that was referred
Feasibility of recruitment and enrollment to study: number of participants enrolled | Screening and baseline
  Tracking number of participants that enrolled into the study
Feasibility of recruitment and enrollment to study: reasons for non-participation | Screening and baseline
  Tracking number of participants who did not enroll into the study and any reasons given by these participants
Adoption outcome: group attendance | During intervention, post-intervention (after 8 weeks of intervention)
  Tracking group attendance per session
Adoption outcome: group completion | During intervention, post-intervention (after 8 weeks of intervention)
  Tracking how many participants completed the group
Adoption outcome: reasons for non-completion | During intervention, post-intervention (after 8 weeks of intervention)
  Tracking the reasons why participants did not complete the group
Acceptability outcome | Post-intervention (after 8 weeks of intervention), and at 3-month follow-up
  Determining the acceptability of the program among participants and facilitators via questionnaires about their experience in the program.
Adherence with intervention protocol: therapist adherence | During and post-intervention (after 8 weeks of intervention)
  (1) assessing therapist adherence to ACT-PM intervention via self-report from therapists and (2) independent rater review of 10% of audio tapes of sessions using ACT-FM (The ACT Fidelity Measure)
Adherence with intervention protocol: completion of participant questionnaires | Baseline, during intervention, post-intervention (after 8 weeks of intervention), and at 3-month follow-up
  Tracking number of participants who completed data collection measures (i.e.. acceptability questionnaire, and clinical scales - described below)

SECONDARY OUTCOMES:
Exploratory clinical symptoms outcome: McMaster Premenstrual And Mood Symptom Scale (MAC PMSS) | Baseline, post-intervention (after 8 weeks of intervention), and at 3-month follow-up
  Individuals can track their mood and premenstrual symptoms on a daily basis using the validated and self-reported McMaster Premenstrual And Mood Symptom Scale (MAC PMSS). The MAC PMSS consists of two charts 1) mood symptom chart, 2) premenstrual symptom chart with severity scores ranging from 1 (not at all) to 6 (extreme). Higher scores indicate a worse outcome.
Exploratory clinical symptoms outcome: Premenstrual Symptoms Screening Tool (PSST) | Baseline, post-intervention (after 8 weeks of intervention), and at 3-month follow-up
  Premenstrual Symptoms Screening Tool (PSST) is a validated questionnaire which consists of 19 questions regarding how symptoms interfere with relationships and daily activities -14 questions are related to premenstrual symptoms, and 5 questions that measure the severity of interference of the symptoms on a woman's ability to function. The scale of each item ranges 0-3: not at all (0); mild (1); moderate (2); severe (3). Higher scores indicate a worse outcome.
Exploratory clinical symptoms outcome: The Patient Health Questionnaire-9 (PHQ-9) | Baseline, post-intervention (after 8 weeks of intervention), and at 3-month follow-up
  9-item assessment for depression, with scores indicating how often symptoms are bothersome, ranging from 0 (not at all) to 3 (nearly every day). Higher scores indicate a worse outcome.
Exploratory clinical symptoms outcome: The Generalized Anxiety Disorder-7 (GAD-7) | Baseline, post-intervention (after 8 weeks of intervention), and at 3-month follow-up
  The GAD-7 a 7-item well-validated self-report scale which can aid in diagnosis and severity assessment for anxiety disorders (including GAD, social anxiety disorder, post-traumatic stress disorder, panic disorder). It is sensitive to change across treatment. Score ranges are from 0-21, with scores of 0-4 representing minimal, 5-9 mild, 10-14 moderate, and 15-21 severe anxiety symptoms.
Exploratory clinical symptoms outcome: The Acceptance and Action Questionnaire (AAQ-II) | Baseline, post-intervention (after 8 weeks of intervention), and at 3-month follow-up
  The AAQ-II is a 7-item self-report scale that assesses constructs relating to acceptance, experiential avoidance, and psychological inflexibility, which are targets of Acceptance and Commitment Therapy (ACT). It has demonstrated satisfactory reliability and validity, has been validated in psychiatric populations, and scores are predictive of mental health and functional outcomes. Higher scores indicate less (worse) flexibility.
Exploratory clinical symptoms outcome: The Mindfulness Attention Awareness Scale (MAAS) | Baseline, post-intervention (after 8 weeks of intervention), and at 3-month follow-up
  The MAAS is a 15-item self-report scale-used previously in both ACT and PMS research-to assess components of mindfulness such as present-moment awareness and observing capacity, which are considered transdiagnostic processes underlying various forms of psychopathology. Higher scores indicate less mindfulness (worse).
Exploratory clinical symptoms outcome: The Valuing Questionnaire (VQ) | Baseline, post-intervention (after 8 weeks of intervention), and at 3-month follow-up
  The VQ is a 10-item self-report measure that was developed to assess changes in a target of ACT-valued living. Its' 2 subscales are correlated strongly with measures of emotional/affective symptoms and life satisfaction. In scoring, higher scores on the Progress scale are associated with health, as are lower scores on the Obstruction scale.
Exploratory clinical symptoms outcome: The Emotion Regulation Questionnaire (ERQ). | Baseline, post-intervention (after 8 weeks of intervention), and at 3-month follow-up
  The ERQ is a 10-item self-report measure designed to assess individuals' tendency to regulate their emotions through Cognitive Reappraisal and Expressive Suppression. Emotion regulation is a target in ACT therapy. To score the ERQ, the average of the scores in each subscale - (i) cognitive reappraisal and (ii) expressive suppression are taken. The higher the score, the greater the use of that particular emotion regulation strategy - cognitive reappraisal is considered adaptive (thus higher scores are better) and expressive suppression maladaptive (lower scores are better).

CONTACTS AND LOCATIONS:
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No